CLINICAL TRIAL: NCT02534441
Title: Epidemiology and Co-Reactivity of Novel Surfactant Allergens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Erin Warshaw, M.D., M.S., Minneapolis Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 4596-A
Record Dates: First submitted 2015-08-06; First posted 2015-08-27 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Allergic Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — Patch Tests

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Skin patch testing to 6 known and 3 novel surfactants (Experimental)
  Interventions: Other: Skin patch test

INTERVENTIONS:
Other: Skin patch test

SUMMARY:
The primary objectives of this study are to identify positivity rates to three novel surfactants (ingredients used in soaps, detergents, and other cleansers that serve to lower the surface tension of the skin and remove debris) and co-reactivity with other surfactants in patients with known surfactant sensitivity on skin patch testing. The investigators hypothesize that subjects who previously tested positive to known allergenic surfactants (cocamidopropyl betaine, stearamidopropyl dimethylamine, dimethylaminopropylamine, coconut diethanolamide, oleamidopropyl dimethylamine, and decyl glucoside) may demonstrate co-reactivity to the three novel surfactant sensitizers (sodium lauroyl sarcosinate, isostearmidopropyl morpholine lactate, and disodium lauroamphodiacetate) on skin patch testing.

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of a previous contact allergy to one or more surfactant(s) on our screening series including:

   * cocamidopropyl betaine
   * stearamidopropyl dimethylamine
   * dimethylaminopropylamine
   * coconut diethanolamide
   * oleamidopropyl dimethylamine, and
   * decyl glucoside
2. Age 18 years or greater.

Exclusion Criteria:

1. Pregnant or lactating women
2. Use of systemic therapy (corticosteroid, immunosuppressive agents, cytostatics, pentoxifylline, leukotriene antagonists or other medication known or suspected to have an effect of ACD) within two weeks prior to participation
3. Use of intramuscular steroids in the last month.
4. Phototherapy (PUVA or UVB) within two weeks prior to participation.
5. Direct sunlight or tanning booth use to the back within the two weeks prior to participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with positive skin patch test reaction, scored using the North American Contact Dermatitis Group (NACDG) criteria, to three novel surfactant antigens. | Five days
  NACDG Scoring as follows: 6=no reaction, 4=doubtful (faint erythema with no induration), 1= mild (erythema, induration, +/- papules), 2=moderate (erythema, induration, papules, vesicles), 3=severe (intense erythema, induration, coalescing vesicles, bullae, spreading), and 5= irritant.